CLINICAL TRIAL: NCT00485407
Title: Guiding Dose Increases In Patients Incompletely Responsive to Usual Doses of Atomoxetine by Determining Plasma Atomoxetine Concentrations: a Randomized, Double-Blind Study
Brief Title: Guiding Dose Increases in Patients Incompletely Responsive to Usual Doses of Atomoxetine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8226; B4Z-MC-LYCL
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

INTERVENTIONS:
Drug: Atomoxetine Hydrochloride

SUMMARY:
The purpose of this trial is to test the value of dose increases in patients with residual ADHD symptoms after treatment with the usual target dose of atomoxetine

ELIGIBILITY:
Inclusion Criteria:

* Outpatients who are at least 6 years of age and not more than 16 years of age at Visit 1
* Patients must meet DSM-IV diagnostic criteria for ADHD (any subtype)
* Patients must have laboratory results showing no significant abnormalities (significant would include laboratory deviations requiring acute medical intervention or further medical evaluation)
* Patients must be of normal intelligence as assessed by the investigator (that is, without a general impairment of intelligence and likely, in the investigator's judgment, to achieve a score of greater than or equal to 70 on an IQ test)
* Patients must be able to swallow capsules

Exclusion Criteria:

* Patients who weigh less than 25 kg or greater than 70 kg at study entry
* Patients with current or past Bipolar I or II disorder, psychosis, autism, Asperger's syndrome, or pervasive developmental disorder
* Patients with a history of any seizure disorder (other than febrile seizures) or patients who have taken (or are currently taking) anticonvulsants for seizure control
* Patients with a history of severe allergies to more than 1 class of medications or multiple adverse drug reactions
* Patients with cardiovascular disease or other conditions that could be aggravated by an increased heart rate or increased blood pressure

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 377 (Actual)
Dates: Start 2003-07; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Test whether patients treated with atomoxetine 1.2 mg/kg/day who have sub-optimal clinical responses and peak plasma atomoxetine levels no higher than 800 ng/mL will benefit from a dose increase to 2.4 mg/kg/day

SECONDARY OUTCOMES:
Assess the relationship between plasma atomoxetine concentration levels and ADHD symptom response
Compare the efficacy of atomoxetine up to 2.4 mg/kg/day with atomoxetine at 1.2 mg/kg/day in reducing residual ADHD symptoms
Assess the safety and tolerability of atomoxetine at doses up to 2.4 mg/kg/day compared to 1.2 mg/kg/day in patients with peak plasma atomoxetine concentration levels no higher than 800 ng/mL as assessed by AEs elicited during open-ended questioning

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scottsdale, Arizona, United States
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, British Columbia, Canada

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com